CLINICAL TRIAL: NCT04038528
Title: Effect on Glucose Control and Quality of Life for People With Type 2 Diabetes of Using a Device to Measure Glucose Levels at Home and Send Them to the Clinic, Rather Than Attending an Out-patient Clinic for Blood Tests
Brief Title: Telemedical Devices in the Management of Type 2 Diabetes Mellitus to Improve Diabetic Control and Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro Studi Internazionali, Italy (Network)
Collaborators: GPI SpA (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-DC-2-0
Record Dates: First submitted 2019-07-23; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telemedicine Group: Patients in this group monitor blood sugar levels at home and upload their data through a telemedicine systems.
  Interventions: Behavioral: telemonitoring of T2DM
- Control Group: The control group will attend their routine appointments scheduled by their GPs and specialists in outpatient clinics and will record blood sugar levels according to the traditional method as per GP or specialist physician's indications.

INTERVENTIONS:
Behavioral: telemonitoring of T2DM — Baseline record of:
  * Weight
  * Height
  * BMI
  * Abdominal circumference
  * Winsor Index
  * ECG
  * Retinography
  * Blood level of (fasting values): total cholesterol, HDL cholesterol, LDL cholesterol, blood sugar, triglycerides, glycated hemoglobin These parameters will be checked again at 3, 6 and 18 months in the two groups.
  Telemedicine group (intervention):
  * Blood sugar (two measurements per week).
  * Body weight (weekly)
  * Blood pressure (weekly) Use of devices that allow the automatic upload of data via wi-fi or web is allowed
  Control group (control):
  Routine appointments scheduled by their GPs and specialists in outpatient clinics to record blood sugar levels as per standard GP or specialist physician's indications.
  Blood sugar level is measured in mg/dl in a drop of capillary blood with the use of standard glucose meter
  Groups: Telemedicine Group

SUMMARY:
The aim of this study is to understand, in adult patients with Type 2 diabetes mellitus, if the use of telemedicine (monitoring and treatment without patients having to attend a healthcare facility) and home-based care is more effective than traditional general practitioner (GP) and outpatient care in terms of patients taking medication regularly and their quality of life.

The hypothesis of this study is that patients with Type 2 diabetes mellitus uploading data on a telemedicine system achieve a glycemic control, evaluated in terms of glycated hemoglobin levels, similar to that of patients followed in a traditional diabetes outpatient department, with improvements to quality of life

DETAILED DESCRIPTION:
Background and study aims Diabetes mellitus is a long-lasting disease in which the level of blood sugar is higher than normal. High level of sugar in the blood can lead to serious consequences, including blindness, kidney failure, amputation of limbs, coma and death. Patients with diabetes need to regularly take their medicine and to make sure they monitor the level of sugar in their blood on daily basis. This can affect their quality of life. The aim of this study is to understand if telemedicine (monitoring and treatment without patients having to attend a healthcare facility) and home-based care is more effective than traditional GP and outpatient care in terms of patients taking medication regularly and their quality of life.

Who can participate? Men and women who live in the study area, have been diagnosed with type 2 diabetes at least 1 year before the start of the study and have been on the same treatment for at least 3 months.

What does the study involve? The participants will be recruited by GPs and doctors working in diabetes centres. Participants will be randomly assigned to one of two groups. One group will be treated and followed according as usual. They will test their blood sugar level at home and record it on paper. They will attend a diabetes outpatient clinic for follow-up. The other group will record the level of blood sugar using a digital home-based system that will send data to the diabetes clinic for follow-up. All participants will receive treatment as appropriate from the clinic. At the end of the study (after 18 months), the two groups will be compared to assess which group achieved a better control of their blood sugar level and which experienced a better quality of life, assessed using a questionnaire. The participants will also have their height, weight, waist circumference, blood pressure, cholesterol and blood fats measured at the beginning and end of the study.

What are the possible benefits and risks of participating? All patients will receive medication as usual and the control group will continue to attend outpatient clinic, so there are no additional risks associated with participating in the trial. The telemedicine group might benefit from avoiding the inconvenience of having to attend outpatient clinics and from a more rapid response to changes in their blood sugar level from the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus (T2DM)
2. Diagnosis of DM made at least 1 year before the start of the study
3. Hypoglycemic treatment remained the same in the 3 months preceding the start of the study

Exclusion Criteria:

1. Diabetes other than T2DM
2. Pregnant women
3. Chronic conditions other than T2DM
4. Unable to give informed consent
5. Dementia or psychiatric conditions that can affect a person's will or ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 2 diabetes mellitus (T2DM) with diagnosis of DM made at least 1 year before the start of the study
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
glycated hemoglobin (GlyH) level | 18 months
  Level of glycated hemoglobin (GlyH) at the end of the study (18 months) in patients followed with telemedicine and in the control group when compared to baseline, with normal GlyH defined as <5.6%.

SECONDARY OUTCOMES:
Quality of life perception | 18 months
  Quality of life as perceived by the patients measured using the SF-36 questionnaire at baseline, 6 months and at the end of the study (18 months)
Body mass index (BMI) | 18 months
  BMI calculated from height and weight at baseline and at the end of the study
Abdominal circumference | 18 months
  Difference in the abdominal circumference measured at baseline and at the end of the study
Triglyceride | 18 months
  Blood triglyceride level at baseline and at the end of the study
LDL-cholesterol | 18 months
  Blood LDL-cholesterol level at baseline and at the end of the study
Systolic Blood Pressure (BP) | 18 months
  Systolic BP at baseline and at the end of the study
Diastolic BP | 18 months
  Diastolic blood pressure at baseline and at the end of the study
Compliance | 18 months
  Compliance with blood glucose testing (number of actual measurements/expected number of measurements in the whole timeframe of the study), with participants divided into four groups: poor (<50%), mediocre (50-70%), good (70-90%), optimal (90-100%)
Hyperglycemic events | 18 months
  Number of hyperglycemic events during the timeframe of the testing, defined as a spot measure of fasting blood sugar >300 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Antonio V Gaddi, MD, PhD, Principal Investigator — EuroGenLab, Bologna, Italy
Locations (1):
- ASP Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be available upon request from DIGITCAL (digitcal01@gmail.com). Anonymised data will be made available to recognised research institutions for research purposes. Written request is required, and data will be shared after approval of the scientific and ethical committees of DIGITCAL. Criteria for data sharing are under discussion at the moment.
Time Frame: Not decided yet
Access Criteria: Not decided yet